CLINICAL TRIAL: NCT01642160
Title: ICAN (Improvement in CPAP Adherence Via the Net) Study
Brief Title: Continous Positive Airway Pressure (CPAP) Compliance Study
Acronym: ICAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, John G. Park, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-008195
Record Dates: First submitted 2012-07-13; First posted 2012-07-17 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of care (Active Comparator): Participants randomized to this arm will have the usual follow up care without any additional information.
  Interventions: Behavioral: Standard of care
- Additional Education (Active Comparator): This arm will receive a weekly text message or e-mail asking participants to sign on to the web page that we will provide. Once they sign on, they will see additional educational materials and questions regarding their CPAP use. Based on their response, they will be directed to suggestion or sites to help improve their compliance with their CPAP.
  Interventions: Behavioral: additional educational material

INTERVENTIONS:
Behavioral: additional educational material — The internet-based intervention group would receive a weekly text or an email (based on the subject's preference). The content of the message asks about their approximate compliance over the past week. Based on their response, they will be directed to one of two internet web pages.
  Arms: Additional Education
Behavioral: Standard of care — participants will receive education from staff nurses as needed.
  Arms: Standard of care

SUMMARY:
Does an internet based text or email interaction and education improve CPAP compliance for patients with Obstructive sleep apnea (OSA) and reduce nursing intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 18 - 90 years of age) newly diagnosed with OSA who have been recommended CPAP therapy.

Exclusion Criteria:

* Previously attempted CPAP, requires the use of bilevel positive airway pressure device, difficulty with English language such that they have difficulty understanding instructions given at high school equivalent, periodic limb movement associated arousals greater than 20/hour, primary complaint of insomnia, diagnosis of restless leg syndrome or periodic limb movement disorder

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
change in mean number of nursing interventions at one month | baseline to one month after initiation

CONTACTS AND LOCATIONS:
Overall Officials: John Park, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States